CLINICAL TRIAL: NCT00003781
Title: Phase II Study of Weekly Docetaxel (Taxotere) in Hormone Refractory Metastatic Prostate Cancer
Brief Title: Docetaxel in Treating Patients With Stage IV Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Purpose: Treatment
Other Study IDs: CDR0000066913; OHSU-5134; OCC-HOR-98037-L; RP-OHSU-5134; NCI-V99-1519
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Pain; Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer; pain
MeSH Terms: conditions — Pain; Prostatic Neoplasms | interventions — Docetaxel; Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: docetaxel
Procedure: pain therapy
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial of docetaxel in treating patients who have stage IV prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of weekly docetaxel as measured by disease response, strength and duration of pain reduction, and either a decrease in analgesic use without an increase in pain, or a decrease in PSA, in patients with hormone refractory metastatic prostate cancer. II. Assess the efficacy of this regimen in terms of survival in this patient population. III. Evaluate the effect of this regimen on quality of life in these patients. IV. Determine qualitative and quantitative toxicities of this regimen in these patients.

OUTLINE: Patients receive docetaxel IV over 15-30 minutes weekly for 6 weeks. Courses repeat every 8 weeks. Therapy continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at weeks 1, 3, 5, and 7 of each course, and a daily pain medication diary is maintained during treatment. Patients are followed for 1 month or until resolution of toxicity, then every 3 months until death.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IV hormone refractory adenocarcinoma of the prostate Symptoms and evidence of disease progression despite standard hormonal therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: At least 3 months Hematopoietic: WBC at least 3000/mm3 Neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) ALT no greater than 2 times ULN (no greater than 1.5 times ULN if alkaline phosphatase is greater than 2.5 times ULN) Alkaline phosphatase no greater than 4 times ULN (no greater than 8 times ULN if known bone involvement and bilirubin and ALT in normal range) Renal: Not specified Other: At least 5 years since any prior malignancy except nonmelanoma skin cancer No other significant medical illness that would prevent compliance No hypersensitivity to drugs formulated with polysorbate-80 Must be able to complete written questionnaires and diaries

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: At least 1 month since prior radiotherapy At least 2 months since prior strontium-89 Surgery: Not specified Other: At least one month since prior investigational agents

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1998-12; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Beer, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States